CLINICAL TRIAL: NCT03138369
Title: Vestibular Stimulation To Trigger Adipose Loss (Vestal) Clinical Trial
Brief Title: Vestibular Stimulation to Trigger Adipose Loss Clinical Trial
Acronym: VeSTAL
Status: Terminated | Type: Interventional
Why Stopped: High drop out rate due to subjects needing to record details of every meal
Sponsor: Neurovalens Ltd. (Industry)
Collaborators: University of California, San Diego (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 170255
Record Dates: First submitted 2017-04-24; First posted 2017-05-03 (Actual); Results first posted 2022-04-27 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-03

CONDITIONS: Obesity; Obesity, Abdominal; Metabolic Syndrome; Weight Loss
Keywords: Obesity; Metabolic Syndrome; Prediabetes; Glycemic control; Hypercholesterolemia; Abdominal obesity; Weight Loss
MeSH Terms: conditions — Obesity; Obesity, Abdominal; Metabolic Syndrome; Weight Loss; Prediabetic State; Hypercholesterolemia

STUDY DESIGN:
Intervention Model Description: Parallel Assignment in 1:1 active to control allocation
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blind
Oversight: Data Monitoring Committee: No | Unapproved Device: Yes

ARMS (2):
- Vestibular nerve stimulation (Experimental): Usage of wearable vestibular nerve stimulator that non-invasively stimulates the vestibular nerves by administering a small electrical current through the skin behind the ears. Should be worn up to one hour a day and at least 5 hours a week.
  Interventions: Device: Vestibular nerve stimulator
- Sham vestibular nerve stimulation (Sham Comparator): Usage of wearable control device that appears identical to active device. Instead of stimulating the vestibular nerves this device will discharge its battery into an internal resistor. Should be worn up to one hour a day and at least 5 hours a week.
  Interventions: Device: Sham vestibular stimulation

INTERVENTIONS:
Device: Vestibular nerve stimulator — Battery powered headset that can be recharged when not being used.
  Other Names: Galvanic vestibular stimulation
  Arms: Vestibular nerve stimulation
Device: Sham vestibular stimulation — Identical in external appearance to the vestibular nerve stimulation device, this device is also powered by a battery and needs to be periodically recharge when not being used. However it discharges into an internal resistor and does not stimulate the vestibular nerve.
  Arms: Sham vestibular nerve stimulation

SUMMARY:
There is an ongoing and worsening problem with obesity in the developed, and much of the developing world. Although it has long been realized that Western diets that are rich in sugar and fat play an important role in this, it has only recently been realized that exposure to these diets, particularly in childhood, can damage the part of the brain that determines how much fat there is in the body. The result of this damage is that the so-called "set-point" for fat in this part of the brain is pushed upwards. There is a lot of evidence from animals that activating the brain's balance (vestibular) system pushes this set-point for fat downwards to cause fat loss, probably because this tricks the brain into thinking that the animal is more physically active. The aim of this study is to see whether the same effect can be triggered in humans by non-invasively stimulating the vestibular system with a small electrical current through the skin behind their ears.

DETAILED DESCRIPTION:
There is a growing realization that obesity can, in many ways, be viewed as a neurological disease triggered by lifestyle factors. There is clear evidence that the arcuate nucleus in the hypothalamus regulates a "set-point" for how much fat the body should have. It does so by altering appetite and metabolic rate so that deviations too far in either direction are strongly resisted. This set-point is determined by genetic, epigenetic and lifestyle factors. Thus, excessive exposure to dietary monosaccharides, such as glucose, and saturated fats, especially in childhood and adolescence, can damage the neurons of the arcuate nucleus and push the set-point up. This then can condemn sufferers to a lifetime of obesity.

Establishing a method of tuning down the set-point for body fat thus has to be a goal if we are to successfully combat the current obesity pandemic. A significant amount of animal work suggests that stimulating the vestibular system in the inner ear, by means of chronic centrifugation, actually does just that and causes a reduction in body fat. This is likely because the chronic vestibular activation is taken by the brain to represent a state of increased physical activity, and in order to optimize homeostasis it would be appropriate for the body to have a leaner physique, by reducing unnecessary energy expenditure from carrying excess fat.

It is possible to stimulate the vestibular nerve in humans by applying a small electrical current to the skin behind the ears. This is an established technology that is believed to be safe, but only previously used for research purposes. We found in a pilot study that recurrent stimulation of this kind for two or three hours a week over four months led to a statistically significant reduction in truncal fat in the active group as opposed to the control group who underwent sham stimulation.

Given the current, and increasing levels of global obesity, it is important to determine whether non-invasive electrical vestibular nerve stimulation (VeNS), otherwise known as galvanic vestibular stimulation, is a viable treatment option. Changes in body fat will be measured using dual energy X-ray absorptiometry (DEXA) scans.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent

   Body mass index (BMI) ≥ 30 kg/m2, or BMI ≥ 27 kg/m2 with one or more of these obesity related co-morbid conditions:
   1. History of treatment for systemic hypertension
   2. History of treatment for dyslipidemia
   3. History of treatment for sleep apnea syndrome
   4. Stable cardiovascular disease (no change in medication and no active events within 1 year).
2. Males or Females. Note females of child-bearing potential must have a negative urine pregnancy test at screen and also just before each DXA scan. (As DXA involves a small dose of ionizing radiation). They should agree to follow a physician-approved contraceptive regimen for the duration of the study period (other than DMPA injections as this causes weight gain).
3. 22-80 years of age inclusive on starting the study.
4. Ability and willingness to complete all study visits and procedures.
5. Owner of a smart phone (iOS or Android) in order to access the diet monitoring and advice app, activity monitoring app, and the app that reports on the status of the stimulation devices used in the study.
6. Agreement not to use of prescription drug therapy or the use of over-the-counter weight loss preparations for the duration of the trial.
7. Agreement not to start smoking tobacco or marijuana for the duration of the study.

Exclusion Criteria:

1. History of vestibular dysfunction.
2. History of bariatric surgery, fundoplication, gastric resection or major upper-abdominal surgery (acceptable surgeries include cholecystectomy, hysterectomy).
3. History of skin breakdown, eczema or other dermatological condition (e.g. psoriasis) affecting the skin behind the ears, or of the head and neck.
4. History of weight loss device implantation (e.g. VBloc Maestro or Abiliti), or use of a non-invasive device.
5. Untreated thyroid disorder (stable treatment for 3 months is acceptable).
6. Other endocrinological causes of weight gain (e.g. Cushing's disease, Cushing's syndrome or acromegaly)
7. Previous diagnosis of HIV infection or AIDS (HIV is known to cause a vestibular neuropathy which would prevent VeNS from working).
8. History of cirrhosis, or liver, kidney or heart failure.
9. Chronic pancreatitis.
10. Treatment with prescription weight-loss drug therapy in the year before starting the study.
11. Tobacco or marijuana smoking in the year prior to starting and for the duration of the study.
12. Known genetic cause of obesity (e.g., Prader-Willi Syndrome).
13. Body weight change of more than 10% in either direction within the previous year.
14. Physician-prescribed diet, and/ or current, active member of an organized weight loss program (e.g., Weight Watchers). (Note: study subjects may continue any personal eating plan they were on prior to study enrollment)
15. Diabetes mellitus (Types 1 & 2). (See Section 9 Research Design and Methods, Appendix 3)
16. Diagnosis of epilepsy or use of anti-epileptic medication within six months of starting the study (e.g. for the treatment of peripheral neuropathy)
17. Chronic (more than a month of daily use) treatment with opioid analgesic drugs within the last year.
18. Regular use (more than twice a month) of anti-histamine medication.
19. Use of oral or intravenous corticosteroid medication within a year of starting the study.
20. Use of the beta-blockers atenolol, metoprolol or propranolol within 3 months of starting the study.
21. Current alterations in treatment regimens of anti-depressant medication for whatever reason (other than tricyclic antidepressants) (Note: stable treatment regimen for prior six months acceptable).
22. An active diagnosis of cancer.
23. A myocardial infarction within the preceding year.
24. A history of stroke or severe head injury (as defined by a head injury that required intensive care). (In case this damaged the neurological pathways involved in vestibular stimulation).
25. Presence of permanently implanted battery powered medical device or stimulator (e.g., pacemaker, implanted defibrillator, deep brain stimulator, vagal nerve stimulator etc.).
26. Psychiatric disorders (including untreated severe depression, schizophrenia, substance abuse, bulimia nervosa etc.)
27. Current participant in another weight loss study or other clinical trials.
28. Have a family member who is currently participating or is planning to participate in this study.
29. Subject weighs over 350 pounds as this is the weight limit of the DXA scanner.

Ages: 22 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2017-11-06 (Actual); Primary Completion 2018-12-14 (Actual); Study Completion 2018-12-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Altman Clinical and Translation Research Institute, UC San Diego, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Pilot Study on Biorxiv — http://doi.org/10.1101/087692

RESULTS

PARTICIPANT FLOW:
Groups:
- Sham Vestibular Nerve Stimulation: Usage of wearable control device that appears identical to active device. Instead of stimulating the vestibular nerves this device will discharge its battery into an internal resistor. Should be worn up to one hour a day and at least 5 hours a week.
  Sham vestibular stimulation: Identical in external appearance to the vestibular nerve stimulation device, this device is also powered by a battery and needs to be periodically recharged when not being used. However, it discharges into an internal resistor and does not stimulate the vestibular nerve.
Period: Overall Study
Arm/Group | Vestibular Nerve Stimulation | Sham Vestibular Nerve Stimulation
Started | 11 | 11
Completed | 8 | 3
Not Completed | 3 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vestibular Nerve Stimulation | Sham Vestibular Nerve Stimulation | Total
Number analyzed (Participants) | 11 | 11 | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.4 (12.1) | 59.8 (9.93) | 55.6 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 11 | 19
  Male | 3 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 11 | 11 | 22
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Mean Body Weight (kg)
Description: Mean total body weight loss (TBWL) from the start of treatment (as a percentage of baseline total body weight). Change = 12 month score - baseline score
Time Frame: Baseline and 12 months
Population: Please note this trial was terminated early
Measure: Mean (Standard Deviation); unit: Kilograms (kg)
Arm/Group | Vestibular Nerve Stimulation | Sham Vestibular Nerve Stimulation
Number analyzed (Participants) | 8 | 3
Kilograms (kg) | -1 (6.90) | 2.47 (4.55)

2. Primary Outcome: Change in Categorical Body Weight
Description: Change in Categorical Body Weight measured by BMI:
  Normal: 18.5-24.9 Overweight: 25.0-29.0 Obese: >30.0 Average BMI calculated. Change = 12 month score - baseline score
Time Frame: Baseline and 12 months
Population: Please note this trial was terminated early.
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Vestibular Nerve Stimulation | Sham Vestibular Nerve Stimulation
Number analyzed (Participants) | 8 | 3
kg/m^2 | -0.40 (2.50) | 1.00 (1.83)

3. Secondary Outcome: Visceral Adipose Tissue
Description: The difference in mean percent loss of baseline visceral adipose tissue (in kilograms) in the vestibular stimulation versus sham stimulation group, as measured by means of a whole body DXA scan. Change = 12 month score - baseline score
Time Frame: Baseline and 12 months
Population: Please note this trial was terminated early.
Measure: Mean (Standard Deviation); unit: Grams (g)
Arm/Group | Vestibular Nerve Stimulation | Sham Vestibular Nerve Stimulation
Number analyzed (Participants) | 8 | 3
Grams (g) | -35.9 (106.1) | 172.7 (372.5)

4. Secondary Outcome: Lean Muscle
Description: Change in total lean (muscle) mass in kilograms between vestibular stimulation and sham stimulation groups as assessed using whole body DXA scans.
Time Frame: Baseline and 12 months
Population: Data was not collected
Arm/Group | Vestibular Nerve Stimulation | Sham Vestibular Nerve Stimulation
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Change in Categorical Body Fat
Description: The proportion of subjects who lose at least 5% of baseline total body fat in the active versus placebo treated groups. (As measured by a whole body DXA scan).
Time Frame: Baseline and 12 months
Population: Data was not collected.
Arm/Group | Vestibular Nerve Stimulation | Sham Vestibular Nerve Stimulation
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Change in Mean Body Fat (g)
Description: The difference in mean percent loss of baseline total body fat in the active versus placebo treated groups. (As measured by means of a whole body DXA scan). Change = 12 month score - baseline score
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: Grams (g)
Arm/Group | Vestibular Nerve Stimulation | Sham Vestibular Nerve Stimulation
Number analyzed (Participants) | 8 | 3
Grams (g) | 152.74 (4912.74) | 3769.37 (4651.19)

ADVERSE EVENTS:
Time Frame: 12 months
Description: Low-risk device - Adverse events and serious adverse events were collected throughout the trial and followed-up with, including after trial termination.
Arm/Group | Vestibular Nerve Stimulation | Sham Vestibular Nerve Stimulation
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/11
Serious Adverse Events (participants affected / at risk) | 1/11 | 0/11
Other Adverse Events (participants affected / at risk) | 6/11 | 5/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vestibular Nerve Stimulation (N=11) | Sham Vestibular Nerve Stimulation (N=11)
Multi-resistant bacterial infection - Non-device related SAE (Immune system disorders) | 1 (1) | 0 (0) — Non-device related SAE. Participant required hospitalisation and antibiotics.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vestibular Nerve Stimulation (N=11) | Sham Vestibular Nerve Stimulation (N=11)
Headache (Nervous system disorders) | 4 (4) | 3 (3)
Nausea (Gastrointestinal disorders) | 3 (4) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-30): https://cdn.clinicaltrials.gov/large-docs/69/NCT03138369/Prot_SAP_000.pdf